CLINICAL TRIAL: NCT00030225
Title: Phase 2 Evaluation of the Vitagen Extracorporeal Liver Assist Device (ELAD) System in the Management of the Patients With Fulminant Hepatic Failure
Brief Title: Phase 2 Evaluation of the ELAD System in the Management of Acute Liver Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vital Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-202
Record Dates: First submitted 2002-02-11; First posted 2002-02-12 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Fulminant Hepatic Failure
Keywords: Fulminant Hepatic Failure
MeSH Terms: conditions — Liver Failure, Acute | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ELAD (Experimental): Treatment with ELAD, extracorporeal liver assist system and standard of care
  Interventions: Biological: ELAD
- Standard of care (Control) (Other): Standard of care for patients with fulminant hepatic (liver) failure
  Interventions: Other: Standard of care (Control)

INTERVENTIONS:
Biological: ELAD
  Other Names: Extracorporeal Liver Assist Device
  Arms: ELAD
Other: Standard of care (Control)
  Arms: Standard of care (Control)

SUMMARY:
The purpose of this study is to determine if treatment with the ELAD Bioartificial Liver Assist Device is beneficial to patients in Acute Liver Failure either as a bridge to liver transplant or bridge to native liver recovery.

DETAILED DESCRIPTION:
Current treatment with modalities in Acute Liver Failure still carry unacceptable morbidity and mortality. It is hoped that by intervening with ELAD a patient will have an opportunity to be bridged to transplant or to avoid transplantation and to have their native liver recover.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of Fulminant Hepatic Failure with encephalopathy, and coagulopathy
* Weight not less than 40 kilograms
* Not listed for organ transplant, but no medical contraindications for transplant

Exclusion Criteria:

* Listed for organ transplant at stud entry
* History of jaundice for greater than 28 days at screening
* Liver dysfunction due to trauma
* Concomitant serious disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2002-01; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects reaching 30-Day survival | Study Day 30
  30-day survival

SECONDARY OUTCOMES:
30-day transplant-free survival | Study Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Maguire, MD, PhD, Study Chair — VitaGen
Locations (7):
- United States (7):
  - UCSD, San Diego, California
  - University of Miami, Miami, Florida
  - Emory School of Medicine, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Background] Millis M, Maguire P, Cronin D, Conjeevarum H, Johnson R, Conlin C, Brotherton J, O'Laughlin R, Triglia D, Piazza R: Continuous Human Liver Support As A Bridge To Transplantation. Hepatology- Vol.30, No.4 October 1999 p168A.